CLINICAL TRIAL: NCT06402695
Title: Observational Study on Clinical, Laboratory, Anatomopathological and Molecular Characteristics and Their Prognostic and Predictive Value in Patients With Neuroendocrine Tumors of the Gastroenteropancreatic Tract and Pulmonary Treated at Fondazione Policlinico Agostino Gemelli (FPG)-IRCCS
Brief Title: Observational Study on GEP-and Pulm-NET Treated at FPG
Acronym: ETNA-FPG
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5981
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Neuroendocrine Tumors; Gep Net; Pulmonary Neuroendocrine Neoplasm
MeSH Terms: conditions — Neuroendocrine Tumors; Gastro-enteropancreatic neuroendocrine tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective cohort: GEP- and Pulm- NET patients referred to the U.O.C. of Medical Oncology of the FPG - IRCCS since 01/01/2010 up to the date of approval of the study.
- prospective cohort: GEP- and Pulm- NET patients referred to the U.O.C. of Medical Oncology of the FPG - IRCCS starting from the date of approval of the study for the following 36 months.

SUMMARY:
Observational ambispective monocentric study on the clinical, laboratory, pathological and molecular characteristics of patients suffering from gastroenteropancreatic tract and pulmonary neuroendocrine tumors and their prognostic and predictive value.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NETs) are a heterogeneous group of rare epithelial neoplasms arising from cells of the diffuse neuroendocrine system. In recent years their incidence has been constantly increasing and up to 80% of cases already begin in an advanced stage. The most frequent site of primary localization is the gastroenteropancreatic tract (GEP-NET) in 60% of cases, followed, in 25%, by the lung (L-NET). Clinically, NETs are classified as functioning (F) or non-functioning (NF) based on the presence of symptoms caused by hormonal secretion produced by tumor cells. NETs are characterized by great clinical and biological, inter- and intra-tumoral heterogeneity. The WHO classification identifies four categories: well-differentiated NETs, G1, G2 and G3, and poorly differentiated neuroendocrine carcinomas (NECs), which represent 10%-20% of all neuroendocrine neoplasms. This classification, together with the TNM stage according to the American Joint Committee on Cancer (AJCC 8th edition) takes on an important prognostic value. However, these two criteria are not exhaustive in predicting the aggressiveness of the pathology nor the response to oncological therapies. There is therefore a clear clinical need, to date unsatisfied, for new prognostic and predictive biomarkers, which can better define the heterogeneity of NETs by implementing classification and staging, to guide prognosis and support therapeutic decisions.

The main feature of all well-differentiated NETs is the overexpression of the somatostatin receptor, measured by PCR-based or immunohistochemistry (IHC)-based methods or by imaging. Among these receptors, the SSTR2A subtype is the most commonly expressed. Diagnostic and therapeutic approaches aimed at SSTR have shown advantages but it is not clear how much the degree of expression of SSTR in positive patients influences the response to treatment and whether it has a correlation with survival, regardless of the oncological treatments used. Furthermore, since the expression of this receptor appears inversely proportional to the degree of differentiation and can be different within the same disease between primary tumor and metastatic disease, this receptor could have a further role as a measure of tumor heterogeneity and disease progression.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of gastroenteropancreatic or pulmonary NET
* age ≥ 18 years;
* radiological evidence of resectable/locally advanced/metastatic disease;
* signing of informed consent;
* at least one visit following the first oncological visit.

Exclusion Criteria:

* absence of clinical data that allow adequate definition of survival (primary endpoint of the study);
* absence of histological diagnosis;
* failure to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years affected by gastroenteropancreatic or pulmonary NET.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | from randomization to end of study or death event (estimed: up to 36 months).
  The length of time from the date of diagnosis to death.

SECONDARY OUTCOMES:
Progression Free Survival | from randomization to progression or death event or end of the study (estimed: up to 36 months).
  The length of time from the date of diagnosis to disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Schinzari, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli - IRCCS, Rome, Italy